CLINICAL TRIAL: NCT00317863
Title: Zink and Bone Strength
Status: Completed | Type: Observational
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: ON-04-003-JO
Record Dates: First submitted 2006-04-23; First posted 2006-04-25 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Coxarthrosis; Fracture of Femoral Neck
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Zink and bone strength

DETAILED DESCRIPTION:
blood- and urine samples collected from 20 OA patients and 20 osteoporosis patients who all had a hip-replacement. All patients were evaluated by DEXA-scanning.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women with osteoarthrosis or femoral neck-fracture i one hip

Exclusion Criteria:

pathology or prosthesis in contralateral hip

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: blood- and urine samples collected from 20 OA patients and 20 osteoporosis patients who all had a hip-replacement. All patients were evaluated by DEXA-scanning.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2008-01-01 (Actual); Study Completion 2008-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janne Ovesen, MD, Principal Investigator — Northern Orthopaedic Division
Locations (1):
- Northern Orthopaedic Division, Klinik Farsoe, Farsø, Northern Jutland, Denmark

REFERENCES:
- See also: Final publication — http://www.ncbi.nlm.nih.gov/pubmed/18398256?dopt=abstract